CLINICAL TRIAL: NCT01321190
Title: Pain Quality in Individuals With Low Back Pain, Headache, and Fibromyalgia
Brief Title: Pain Quality Study
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mark Jensen, Principal Investigator, University of Washington
Other Study IDs: 40324-EA
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Low Back Pain; Headache; Fibromyalgia
MeSH Terms: conditions — Low Back Pain; Headache; Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Low Back Pain: Individuals who experience bothersome low back pain.
- Headache: Individuals who experience bothersome headaches.
- Fibromyalgia: Individuals who experience bothersome fibromyalgia-related pain.

SUMMARY:
One way to better understand how various treatments for pain differ is to determine the effects of these treatments on different pain qualities or characteristics. For example, pain can be described as "hot", "electrical", "cold", "achy", and "piercing." In order to determine which pain quality/qualities that a pain treatment affects, researchers must develop measures of these pain qualities or characteristics. The purpose of this study is to learn more about the different pain qualities individuals who have low back pain, headaches and fibromyalgia experience. Identifying the common qualities of pain experienced by these groups will help researchers evaluate and develop more comprehensive pain quality measures, which will ultimately help them to be able to test the effectiveness of treatments for these different pain qualities.

ELIGIBILITY:
Inclusion Criteria:

* Speaks and understands English;
* At least 18 years of age;
* Confirms a diagnosis from a physician or certified medical provider of one of the three medical conditions (low back pain, headache, fibromyalgia), and that pain related to this diagnosis is still bothersome.
* Has experienced bothersome pain associated with their diagnosis in the past three months of a sufficient intensity;
* English is their first and primary language.

Exclusion Criteria:

* Individuals would be excluded if they have more than one of the three pain diagnoses to be studied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have a formal diagnosis of one of the three conditions studied and have received services at either or both the Harborview Medical Center and the University of Washington Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pain Quality Assessment Scale | The assessment scale was administered once within a month following enrollment in the study; the assessment scale was not administered within a timeframe specific to an event or onset of condition.
  Assesses qualities (e.g. hot,cold) of pain

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Jensen, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Jensen MP, Johnson LE, Gertz KJ, Galer BS, Gammaitoni AR. The words patients use to describe chronic pain: implications for measuring pain quality. Pain. 2013 Dec;154(12):2722-2728. doi: 10.1016/j.pain.2013.08.003. Epub 2013 Aug 8. PMID 23933183